CLINICAL TRIAL: NCT03753620
Title: Development of a Software Correlating Simultaneously fMRI, EEG and Peripheral Physiological Activity
Acronym: NEUREXPLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: API/2017/91
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Music Listening
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music listening (Experimental): The participants listens to their favorite emotional musical extracts. While listening, their Hemodynamic activity (with fMRI), their cerebral electric activity (with EEG) and their peripheral physiological parameters are recorded simultaneously
  Interventions: Device: simultaneous fMRI and EEG + peripheral measures; Device: EEG and peripheral measures

INTERVENTIONS:
Device: simultaneous fMRI and EEG + peripheral measures — Hemodynamic activity recorded with fMRI, cerebral electric activity recorded with EEG as well as peripheral physiological parameters will be recorded during music listening.
Device: EEG and peripheral measures — cerebral electric( with EEG) as well as peripheral physiological parameters will be recorded during music listening.

SUMMARY:
The study aim to improve the quality of EEG recordings during simultaneous fMRI acquisitions. The second aim is to validate the correspondence between cerebral areas activated in fMRI and cortical areas identified with high density EEG during the listening of emotional musical pieces.

ELIGIBILITY:
Inclusion Criteria:

* Right handed healthy people
* Sensitive to "music chill" (Barcelona Reward music Questionnaire>50)
* Having given their participation agreement
* Individual with health insurance coverage.

Exclusion Criteria:

* Pregnant women
* Individuals in "exclusion period" of another study
* No inclusion criteria of fMRI acquisition
* Subjects with auditory deficits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation between synchronous cerebral hemodynamics and electric patterns recorded with both EEG and fMRI simultaneously during the production of musical emotions. | Day 0
  The cerebral activity will be measured continuously during musical extracts listening and comparison of the participant self report emotional level will allow to compare fMRI and EEG data to ensure a good correspondence.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France